CLINICAL TRIAL: NCT07384598
Title: Pharmacokinetic Profiles of Subcutaneous Enoxaparin for Thromboprophylaxis in Critically Ill Patients With Renal Failure Treated or Not With Continuous Veno-veinous Hemofiltration.
Acronym: AKI-ENOXA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Pierre Ottignies (Other)
Responsible Party: Principal Investigator, Nicolas De Schryver, Principal Investigator, Clinique Saint Pierre Ottignies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AKI-ENOXA
Record Dates: First submitted 2026-01-12; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Thromboprophylaxis; Critical Illness; Intensive Care (ICU)
Keywords: thromboprophylaxis
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thromboprophylaxis arm (Experimental): Participating subjects will be given a prophylactic dose of enoxaparin, via the subcutaneous route, as standard of care. The enoxaparin dose will be defined according to the actual patient's body weight as follow: 40 mg daily for patients between 60 and 100 kg, 30 mg daily for patient < 60 kg and 50 mg daily for patients > 100 kg.
  Interventions: Diagnostic Test: Anti-Xa profiles after the subcutaneous administration of a prophylactic dose of enoxaparin

INTERVENTIONS:
Diagnostic Test: Anti-Xa profiles after the subcutaneous administration of a prophylactic dose of enoxaparin — Monitoring of the antifactor Xa activity will be performed immediately before (H0), 4(H4), 8(H8), 12 (H12), and 24 (H24) hours after up to 3 doses of LMWH administration.

SUMMARY:
Thromboprophylaxis is recommended for critically ill patients without contraindications and is usually achieved by the subcutaneous daily administration of a low dose of low molecular weight heparin (LMWH). The efficacy of this measure can be assessed by measuring the anticoagulation level obtained in the blood by dosing the anti-Xa activity. However, multiple studies have shown that anti-Xa activities in critically ill patients in the intensive care unit (ICU) are much lower, and below the desired range, than their ward counterparts.

LMWH elimination depends on kidney function and reduced dosing is recommended for patients with renal failure, treated or not with renal replacement therapy (continuous veno-venous hemofiltration (CVVH)). However, some scarce data suggest that even critically ill patients with renal failure treated with reduced or even with standard doses of LMWH, also have lower anti-Xa activities (below the desired range). If confirmed, this finding may suggest that reduced or even standard dosing of LMWH for thromboprophylaxis in critically ill patients with renal failure should be replaced by another dosing regimen or another route of administration. Therefore, this study aims to better characterize the pharmacokinetic profiles of LMWH after administration of a prophylactic dose of enoxaparin daily in patients with renal failure treated or not with CVVH, and to compare them to patients with no renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year old
* Hospitalized in the ICU.
* Equiped with an arterial line.
* Indication for thromboprophylaxis with a daily prophylactic dose of enoxaparin.
* Additionnally:

  * For cohort 1: severe renal failure (KDIGO stage ≥2) without CVVH AND SOFA score ≥4.
  * For cohort 2: severe renal failure (KDIGO stage ≥2) with CVVH AND sequential organ failure assessment (SOFA) score ≥4.
  * For cohort 3: no renal failure (creatinine clearance > 60 ml/min)

Exclusion Criteria:

* Platelet count < 50 000/μl.
* CHILD PUGH stage C cirrhosis.
* Known coagulation disorder.
* Patient treated in the last 3 days with direct oral anticoagulants.
* Patient treated in the last 24h with LMWH before enrollment.
* High bleeding risk with contra indication for standard dose of LMWH prophylaxis, as per investigator judgment
* Indication for therapeutic anticoagulation (including CVVH with systemic heparin anticoagulation).
* Body weight < 50 kg or > 120 kg.
* Evidence of recovery of renal function before enrollment, based on investigator judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
mean peak anti-Xa activity | 4 hours after the subcutaneous administration of a prophylactic dose of enoxaparin
  The primary endpoint will be the difference in the mean peak anti-Xa activity 4 hours after the subcutaneous administration of a prophylactic dose of enoxaparin in critically ill patients with renal failure without CVVH (N=20), in patients with renal failure with CVVH (N=20) and in a control group of patients with no renal failure (N=20).

SECONDARY OUTCOMES:
Mean area under the curve (AUC) (0-24 hours) of anti-Xa activity | 0-24 hours after the subcutaneous administration of a prophylactic dose of enoxaparin
Trough value of anti-Xa activity | Trough value of anti-Xa activity 24 hours after the injection of a prophylactic dose of enoxaparin.

IPD SHARING:
Plan to Share IPD: No
There is no intention to share IPD for this trial.